CLINICAL TRIAL: NCT03958006
Title: Simultaneous Cochlear Implantation During Translabyrinthine Resection of Vestibular Schwannoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1349609
Record Dates: First submitted 2019-03-18; First posted 2019-05-21 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Vestibular Schwannoma; Cochlear Implantation
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Cochlear Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cochlear implantation (Experimental): Simultaneous cochlear implantation with tumor resection
  Interventions: Device: Cochlear implant

INTERVENTIONS:
Device: Cochlear implant — Tumor resection with cochlear implant

SUMMARY:
This study will address the feasibility of simultaneous cochlear implantation during resection of a vestibular schwannoma.

DETAILED DESCRIPTION:
This is prospective study patients undergoing a translabyrinthine resection for a vestibular schwannoma with intact hearing in the contralateral ear. During surgery, simultaneous cochlear implantation will be performed if the cochlear nerve can be identified and preserved during the resection.

Relevant data to be collected will include patient demographics, details related to the vestibular schwannoma including side, size, symptoms (specifically pre-operative hearing loss, degree of tinnitus), and status of hearing in the contralateral ear. Surgical details to be recorded will include date of surgery, surgical time, and whether the cochlear nerve was identified and preserved. Details related to the post-operative course to be recorded include length of stay in the hospital, post-operative complications such as wound infection or cerebral spinal fluid (CSF) leak, and need for revision or additional procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a vestibular schwannoma undergoing a translabyrinthine resection with intact hearing in the contralateral ear

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Measurement of Hearing Parameters | 1 month, 3 months and 6 months postoperatively.
  Audiologist assesses changes in understanding of the AzBio test (words in quiet and words in background noise) post cochlear implantation.
Measurement of Hearing Parameters | 1 month, 3 months and 6 months postoperatively.
  Audiologist assesses changes in understanding of 50 random consonant-nucleus-consonant sounds.
Measurement of Hearing Parameters | 1 month, 3 months and 6 months postoperatively.
  Audiologist assesses changes in understanding changes in understanding of Speech, Spatial and Qualities of Hearing.

SECONDARY OUTCOMES:
Measurement of Change of Physical Symptoms Associated with Hearing Loss | 1, 3 and 6 months postoperatively
  Patients will complete the Dizziness Handicap Inventory
Assessment of Change of Physical Symptoms Associated with Hearing Loss | 1, 3 and 6 months postoperatively
  Patients will complete the Tinnitus Handicap Inventory
Assessment of incision site healing | 1 week, and 1 and 3 months postoperatively
  Surgeon evaluates wound hearing over 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Seilish Babu, MD, Principal Investigator — Michigan Ear Institute, Farmington Hills, MI
Locations (1):
- Seilesh Babu, Farmington Hills, Michigan, United States

REFERENCES:
- [Background] Dos Santos Neto PH, Zamponi JO, Hamerschmidt R, Wiemes GRM, Rassi MS, Borba LAB. Simultaneous cochlear implantation as a therapeutic option in vestibular schwannoma surgery: case report. Neurosurg Focus. 2018 Mar;44(3):E9. doi: 10.3171/2017.12.FOCUS17670. PMID 29490548
- [Background] Lloyd SK, Glynn FJ, Rutherford SA, King AT, Mawman DJ, O'Driscoll MP, Evans DG, Ramsden RT, Freeman SR. Ipsilateral cochlear implantation after cochlear nerve preserving vestibular schwannoma surgery in patients with neurofibromatosis type 2. Otol Neurotol. 2014 Jan;35(1):43-51. doi: 10.1097/MAO.0000000000000185. PMID 24335931
- [Background] Bohr C, Muller S, Hornung J, Hoppe U, Iro H. [Hearing restoration with cochlear implants after translabyrinthine vestibular schwannoma resection]. HNO. 2017 Sep;65(9):758-765. doi: 10.1007/s00106-017-0404-2. German. PMID 28819872
- [Background] Hassepass F, Arndt S, Aschendorff A, Laszig R, Wesarg T. Cochlear implantation for hearing rehabilitation in single-sided deafness after translabyrinthine vestibular schwannoma surgery. Eur Arch Otorhinolaryngol. 2016 Sep;273(9):2373-83. doi: 10.1007/s00405-015-3801-8. Epub 2015 Oct 23. PMID 26498948
- [Background] DeHart AN, Broaddus WC, Coelho DH. Translabyrinthine vestibular schwannoma resection with simultaneous cochlear implantation. Cochlear Implants Int. 2017 Sep;18(5):278-284. doi: 10.1080/14670100.2017.1337665. Epub 2017 Jun 12. PMID 28602150
- [Background] Sanna M, Medina MD, Macak A, Rossi G, Sozzi V, Prasad SC. Vestibular Schwannoma Resection with Ipsilateral Simultaneous Cochlear Implantation in Patients with Normal Contralateral Hearing. Audiol Neurootol. 2016;21(5):286-295. doi: 10.1159/000448583. Epub 2016 Nov 5. PMID 27816972
- [Background] Rooth MA, Dillon MT, Brown KD. Prospective Evaluation of Patients Undergoing Translabyrinthine Excision of Vestibular Schwannoma with Concurrent Cochlear Implantation. Otol Neurotol. 2017 Dec;38(10):1512-1516. doi: 10.1097/MAO.0000000000001570. PMID 29099442